CLINICAL TRIAL: NCT05567380
Title: Comparative Study of JAK Inhibitors Vs TNF Inhibitors in Patients With Rheumatoid Arthritis
Brief Title: Comparative Study of Janus Kinase (JAK) Inhibitors Vs Tumor Necrosis Factor (TNF) Inhibitors in Rheumatoid Arthritis
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Esraa Mohamed Mahmoud, Principal Investigator, Sohag University
Other Study IDs: Soh-Med-22-09-06
Record Dates: First submitted 2022-09-22; First posted 2022-10-05 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Rheumatoid Arthritis
Keywords: JAK Inhibitors; TNF Inhibitors
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — Observation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Methotrexate: Patients newly diagnosed with active Rheumatoid Arthritis and receiving lowest effective dosage of Methotrexate as initial therapy.
  Interventions: Other: Observation
- Methotrexate + JAK Inhibitors: Patients diagnosed with active Rheumatoid Arthritis and have shown intolerance or inadequate response to Methotrexate so JAK Inhibitor (Barcitinib) was added at 4mg/day orally to their therapy.
  Interventions: Other: Observation
- Methotrexate + TNF Inhibitors: Patients diagnosed with active rheumatoid arthritis and have shown intolerance or inadequate response to Methotrexate so TNF Inhibitor was added to their therapy (either Golimumab at 50mg subcutaneous injection/m, or Etanercept at 50mg subcutaneous injection/wk)
  Interventions: Other: Observation

INTERVENTIONS:
Other: Observation — Observation of Rheumatoid arthritis disease response to JAK inhibitors and TNF inhibitors after definite timepoints from the initialization of treatment in comparison to the current standard of care of therapy with conventional DMARDs.

SUMMARY:
Rheumatoid arthritis is a systemic autoimmune disease characterized by inflammatory synovitis and progressive joint destruction, which are associated with severe disability and increased mortality. It occurs at an incidence of 5 per 1000 with Women being 2 times more likely to be affected by Rheumatoid Arthritis than men. The peak incidence in both groups is in the sixth decade of life.

Management of RA has improved substantially in recent years. In addition to the reduction of signs and symptoms, improvement of physical function, and inhibition of structural damage, better patient outcomes, and clinical remission are now considered achievable goals. Therefore, the current recommended primary target for the treatment of RA should be a state of clinical remission.

Methotrexate (MTX) should be initiated, typically as monotherapy. If treatment response is inadequate, other Disease-modifying antirheumatic drugs (DMARDs) may be added to (rather than replacing) methotrexate to enhance efficacy and reduce the potential for the formation of anti-drug antibodies. TNF inhibitors are the first-line biologic therapies used in the event of incomplete response or adverse reaction to conventional DMARDs as TNF alpha is an important proinflammatory cytokine produced by macrophages and other cells, with myriad actions relevant to the pathogenesis of RA, including stimulation of other proinflammatory cytokine production, expression of endothelial cell adhesion molecules, production of metalloproteinases, and stimulation of osteoclasts. Activated Janus kinases (JAKs) play pivotal roles in intracellular signaling from cell-surface receptors for multiple cytokines implicated in the pathologic processes of rheumatoid arthritis. Baricitinib, an orally available small molecule, provides reversible inhibition of Janus Kinase 1 (JAK1) and Janus Kinase 2 (JAK2) and has shown clinical efficacy in studies involving patients with moderate to severely active Rheumatoid Arthritis who are either intolerant to MTX treatment or who have had an inadequate response to DMARDs, either conventional or biologic.

DETAILED DESCRIPTION:
Aims of the Study:

* To determine the outcome of patients with moderate to severely active rheumatoid arthritis (RA) - despite methotrexate treatment - on JAK inhibitors (Baricitinib).
* To determine the outcome of patients with moderate to severely active rheumatoid arthritis (RA) - despite methotrexate treatment- on TNF inhibitors (Golimumab and Etanercept).
* To compare the outcome between these 2 groups of patients in terms of improvements in signs and symptoms, physical function, patient-reported outcomes, and progression of structural joint damage.
* Detection of any adverse effects that may emerge during the course of treatment.

Patients will be classified into 3 groups:

group (1): patients receiving Methotrexate group (2): patients receiving Methotrexate in addition to JAK inhibitors (Baricitinib at 4 mg once daily by oral route) group (3): patients receiving Methotrexate in addition to TNF inhibitors (Golimumab at 50 mg/month or Etanercept at 50mg/ week by subcutaneous injections)

ELIGIBILITY:
Inclusion Criteria:

* Age: patients >18 years old.
* Patients with Rheumatoid arthritis diagnosed according to the 2010 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology Classification Criteria for RA.
* Patients with moderate to severely active RA as evaluated by DAS28-Score, who have never been treated with biologic DMARDs and who expressed a lack of adequate response or intolerability to conventional DMARDs.

Exclusion Criteria:

* Age < 18 years.
* Any autoimmune disease other than Rheumatoid arthritis.
* Previous treatment with biologic DMARDs.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will include all patients presented to the Rheumatology department-Sohag University Hospitals from October 1st , 2022 till June 30th , 2023, and were diagnosed with Rheumatoid Arthritis according to the 2010 American College of Rheumatology (ACR)/European Alliance of Associations for Rheumatology Classification Criteria for RA and received conventional DMARDs, TNF inhibitors (Golimumab or Etanercept) or JAK inhibitors (Barcitinib).
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Assessment of TJC and SJC | Change from baseline number of tender and swollen joint count at 6 months
  Assessment of Tender Joints Count (TJC) and Swollen Joints Count (SJC), both are parameters to describe disease severity.
Assessment of Visual Analogue Scale (VAS) | Change from baseline Visual Analogue Scale (VAS) at 6 months
  A patient is asked to indicate his/her perceived pain intensity along a 100 mm horizontal line, and this rating is then measured from the left edge. Minimum score is zero indicating no pain, while maximum score is 100 indicating severe pain.
Assessment of disease activity by DAS28 (Disease Activity Score for 28 Joints) | Change from baseline Disease Activity score for 28 joint (DAS28) at 6 months
  DAS28 (Disease Activity Score for 28 Joints) is a widely used scoring system for assessment of disease activity in Rheumatoid Arthritis patients. Minimum value is zero, which indicates disease remission while maximum value is 9.4, which indicates highest disease activity.
Clinical Disease Activity Index (CDAI) score. | Change from baseline Clinical Disease Activity Index at 6 months
  CDAI score is used in routine assessment of disease activity in RA patients. Minimum score is 0 indicating disease remission , while maximum score is 600 indicating highest disease activity.
Structural joint damage | Change from baseline structural joint damage as measured by Larsen Scoring System at 6 months
  measured by the modified Larsen scoring system using plain x-rays (AP view) on both hands and feet. Minimum score is zero indicating normal joint, while maximum score is 5 indicating complete joint deformation.

CONTACTS AND LOCATIONS:
Overall Officials: Esraa Mahmoud, MBBCh, Principal Investigator — Sohag University

IPD SHARING:
Plan to Share IPD: No
Individual Participant Data (IPD) will not be shared with anyone as per consent

REFERENCES:
- [Background] Smolen JS, Aletaha D, Koeller M, Weisman MH, Emery P. New therapies for treatment of rheumatoid arthritis. Lancet. 2007 Dec 1;370(9602):1861-74. doi: 10.1016/S0140-6736(07)60784-3. PMID 17570481
- [Background] Myasoedova E, Crowson CS, Kremers HM, Therneau TM, Gabriel SE. Is the incidence of rheumatoid arthritis rising?: results from Olmsted County, Minnesota, 1955-2007. Arthritis Rheum. 2010 Jun;62(6):1576-82. doi: 10.1002/art.27425. PMID 20191579
- [Background] Aletaha D, Smolen JS. Diagnosis and Management of Rheumatoid Arthritis: A Review. JAMA. 2018 Oct 2;320(13):1360-1372. doi: 10.1001/jama.2018.13103. PMID 30285183
- [Background] Ting YT, Petersen J, Ramarathinam SH, Scally SW, Loh KL, Thomas R, Suri A, Baker DG, Purcell AW, Reid HH, Rossjohn J. The interplay between citrullination and HLA-DRB1 polymorphism in shaping peptide binding hierarchies in rheumatoid arthritis. J Biol Chem. 2018 Mar 2;293(9):3236-3251. doi: 10.1074/jbc.RA117.001013. Epub 2018 Jan 9. PMID 29317506
- [Background] O'Shea JJ, Kontzias A, Yamaoka K, Tanaka Y, Laurence A. Janus kinase inhibitors in autoimmune diseases. Ann Rheum Dis. 2013 Apr;72 Suppl 2(0 2):ii111-5. doi: 10.1136/annrheumdis-2012-202576. PMID 23532440
- [Background] Kitas GD, Gabriel SE. Cardiovascular disease in rheumatoid arthritis: state of the art and future perspectives. Ann Rheum Dis. 2011 Jan;70(1):8-14. doi: 10.1136/ard.2010.142133. Epub 2010 Nov 24. PMID 21109513
- [Background] Smolen JS, Breedveld FC, Burmester GR, Bykerk V, Dougados M, Emery P, Kvien TK, Navarro-Compan MV, Oliver S, Schoels M, Scholte-Voshaar M, Stamm T, Stoffer M, Takeuchi T, Aletaha D, Andreu JL, Aringer M, Bergman M, Betteridge N, Bijlsma H, Burkhardt H, Cardiel M, Combe B, Durez P, Fonseca JE, Gibofsky A, Gomez-Reino JJ, Graninger W, Hannonen P, Haraoui B, Kouloumas M, Landewe R, Martin-Mola E, Nash P, Ostergaard M, Ostor A, Richards P, Sokka-Isler T, Thorne C, Tzioufas AG, van Vollenhoven R, de Wit M, van der Heijde D. Treating rheumatoid arthritis to target: 2014 update of the recommendations of an international task force. Ann Rheum Dis. 2016 Jan;75(1):3-15. doi: 10.1136/annrheumdis-2015-207524. Epub 2015 May 12. PMID 25969430
- [Background] Singh JA, Saag KG, Bridges SL Jr, Akl EA, Bannuru RR, Sullivan MC, Vaysbrot E, McNaughton C, Osani M, Shmerling RH, Curtis JR, Furst DE, Parks D, Kavanaugh A, O'Dell J, King C, Leong A, Matteson EL, Schousboe JT, Drevlow B, Ginsberg S, Grober J, St Clair EW, Tindall E, Miller AS, McAlindon T; American College of Rheumatology. 2015 American College of Rheumatology Guideline for the Treatment of Rheumatoid Arthritis. Arthritis Care Res (Hoboken). 2016 Jan;68(1):1-25. doi: 10.1002/acr.22783. Epub 2015 Nov 6. PMID 26545825
- [Background] Smolen JS, Landewe R, Breedveld FC, Buch M, Burmester G, Dougados M, Emery P, Gaujoux-Viala C, Gossec L, Nam J, Ramiro S, Winthrop K, de Wit M, Aletaha D, Betteridge N, Bijlsma JW, Boers M, Buttgereit F, Combe B, Cutolo M, Damjanov N, Hazes JM, Kouloumas M, Kvien TK, Mariette X, Pavelka K, van Riel PL, Rubbert-Roth A, Scholte-Voshaar M, Scott DL, Sokka-Isler T, Wong JB, van der Heijde D. EULAR recommendations for the management of rheumatoid arthritis with synthetic and biological disease-modifying antirheumatic drugs: 2013 update. Ann Rheum Dis. 2014 Mar;73(3):492-509. doi: 10.1136/annrheumdis-2013-204573. Epub 2013 Oct 25. PMID 24161836
- [Background] Brennan FM, McInnes IB. Evidence that cytokines play a role in rheumatoid arthritis. J Clin Invest. 2008 Nov;118(11):3537-45. doi: 10.1172/JCI36389. PMID 18982160
- [Background] Burmester GR, Kaeley GS, Kavanaugh AF, Gabay C, MacCarter DK, Nash P, Takeuchi T, Goss SL, Rodila R, Chen K, Kupper H, Kalabic J. Treatment efficacy and methotrexate-related toxicity in patients with rheumatoid arthritis receiving methotrexate in combination with adalimumab. RMD Open. 2017 Sep 17;3(2):e000465. doi: 10.1136/rmdopen-2017-000465. eCollection 2017. PMID 28955494
- [Background] Tanaka Y, Emoto K, Cai Z, Aoki T, Schlichting D, Rooney T, Macias W. Efficacy and Safety of Baricitinib in Japanese Patients with Active Rheumatoid Arthritis Receiving Background Methotrexate Therapy: A 12-week, Double-blind, Randomized Placebo-controlled Study. J Rheumatol. 2016 Mar;43(3):504-11. doi: 10.3899/jrheum.150613. Epub 2016 Feb 1. PMID 26834213
- [Background] Genovese MC, Kremer J, Zamani O, Ludivico C, Krogulec M, Xie L, Beattie SD, Koch AE, Cardillo TE, Rooney TP, Macias WL, de Bono S, Schlichting DE, Smolen JS. Baricitinib in Patients with Refractory Rheumatoid Arthritis. N Engl J Med. 2016 Mar 31;374(13):1243-52. doi: 10.1056/NEJMoa1507247. PMID 27028914
- [Background] Keystone EC, Taylor PC, Drescher E, Schlichting DE, Beattie SD, Berclaz PY, Lee CH, Fidelus-Gort RK, Luchi ME, Rooney TP, Macias WL, Genovese MC. Safety and efficacy of baricitinib at 24 weeks in patients with rheumatoid arthritis who have had an inadequate response to methotrexate. Ann Rheum Dis. 2015 Feb;74(2):333-40. doi: 10.1136/annrheumdis-2014-206478. Epub 2014 Nov 27. PMID 25431052